CLINICAL TRIAL: NCT04907318
Title: Retrospective Study Analysing the Results of Toric and Toric Multifocal Intraocular Lens Implantation During Cataract Surgery.
Brief Title: Comparison Between a Toric Monofocal and Multifocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHY PODT-POD FT
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cataract
Keywords: IOL; Toric; Multifocal
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ANKORIS: Cataract surgery performed with POD26PAYT
  Interventions: Device: Cataract surgery
- FINEVISION TORIC: Cataract surgery performed with POD26PAYFT
  Interventions: Device: Cataract surgery

INTERVENTIONS:
Device: Cataract surgery

SUMMARY:
The primary objective of the study is to observe the rotational stability of the implant 30 minutes, one day, 6 weeks, 6 months and 12 months after the implant surgery. In addition, the refraction will be measured as it is directly affected in the event of postoperative rotation. The correlation between postoperative rotation and the following parameters will be determined: PEXS, white-to-white, age, axial length, anterior chamber depth. Visual acuities with and without correction and the best refraction to assess the benefit of the implants will also be investigated.

DETAILED DESCRIPTION:
This retrospective study will include approximately 90 eyes of patients (adults) receiving conventional cataract surgery having a preoperative corneal astigmatism of 1.0 D or higher. They had been implanted with the Ankoris or T-Flex or FineVision toric implant (about 30/30 and20). So that the groups are comparable, the inclusion and exclusion criteria will be those applicable to a multifocal implant.

Inclusion criteria for research participants.

* Cataract (with or without presbyopia)
* No pre-existing ocular pathology or history of ocular surgery
* No phacodonesis

PEX patients (pseudoexfoliation syndrome) can be included. Exclusion criteria for research participants. To ensure equivalence of the two comparable groups, the patients with potential postoperative visual acuity less than 5/10, particularly due to an insufficient retinal function or poor corneal condition will be excluded.

In particular the patients with the following pathologies will be excluded:

* Irregular astigmatism.
* Cases of uncontrolled glaucoma.
* Intraocular inflammation.
* Narrow anterior chambers (2.5 mm).
* Amblyopia with potential visual acuity less than 5/10.
* Any corneal pathology potentially affecting topography (e.g., keratoconus).
* Patients with a history of corneal surgery (especially refractive surgery).
* Patients with diagnosed degenerative visual disorders (e.g., macular degeneration, diabetic retinopathy or other retina diseases or surgery) with known negative impact on visual function possibly leading to visual acuity levels below 0.5.
* Patients with a history of ocular trauma.
* Pathological miosis.
* Patients with zonular laxity.
* Patients suffering from chronic uveitis.
* Patients with monophthalmia. Capsule rupture, intraocular haemorrhage, excessive loss of vitreous, vitreous flare, soft capsules during cataract surgery are also exclusion criteria.

  3 - Adopted observation or investigation method This study involves the collection of data in patient records that fall within the normal framework of cataract surgery.

The demographic and clinical data collected will be the yeat of birth and patient's gender, including ocular or general comorbidities (such as diabetes or rheumatoid illnesses) justifying the visual acuity performance.

The preoperative data collected will be: visual acuity, intraocular pressure, cell density of the corneal endothelium, axial length and corneal power in both axes (data required to routinely calculate the power of the implant and entered into the record to understand any postoperative refractive errors).

The intraoperative data will be the power of the implant and any complications, if applicable.

The postoperative data will be data collected during the standard postoperative follow-up performed at 30 minutes, 1 day, one week, 6 weeks, 6 months and 1 year, with patient questioning, slit lamp observation with implant position, measuring intraocular pressure, determining the best refraction and measuring visual acuity with and without correction (near, far and intermediate vision).

4 - Origin and nature of collected personal data Reason for using this data Observations will be obtained by the doctor from patient records. Clinical data will be used to link potential poor postoperative visual acuity and a comorbidity.

Refractive data will help determine the implant stability in the eye in terms of its depth, i.e. in the sagittal plane, and its rotational stability, i.e. coronal plane stability.

Changes will determine its stability in the coronal plane around the visual axis.

The intraocular pressure analysis and slit lamp examination will help determine the eye inflammatory status before and after surgery.

The record of postoperative keratometry values will help determine whether the error or a refractive change caused by the corneal instability or by the change in the implant position.

ELIGIBILITY:
Inclusion Criteria:

* Cataract (with or without presbyopia)
* No pre-existing ocular pathology or history of ocular surgery
* No phacodonesis

PEX patients (pseudoexfoliation syndrome) can be included.

Exclusion Criteria:

To ensure equivalence of the two comparable groups, the patients with potential postoperative visual acuity less than 5/10, particularly due to an insufficient retinal function or poor corneal condition will be excluded.

In particular the patients with the following pathologies will be excluded:

* Irregular astigmatism.
* Cases of uncontrolled glaucoma.
* Intraocular inflammation.
* Narrow anterior chambers (2.5 mm).
* Amblyopia with potential visual acuity less than 5/10.
* Any corneal pathology potentially affecting topography (e.g., keratoconus).
* Patients with a history of corneal surgery (especially refractive surgery).
* Patients with diagnosed degenerative visual disorders (e.g., macular degeneration, diabetic retinopathy or other retina diseases or surgery) with known negative impact on visual function possibly leading to visual acuity levels below 0.5.
* Patients with a history of ocular trauma.
* Pathological miosis.
* Patients with zonular laxity.
* Patients suffering from chronic uveitis.
* Patients with monophthalmia. Capsule rupture, intraocular haemorrhage, excessive loss of vitreous, vitreous flare, soft capsules during cataract surgery are also exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This retrospective study will include approximately 90 eyes of patients (adults) receiving conventional cataract surgery having a preoperative corneal astigmatism of 1.0 D or higher and had been implanted with the Ankoris or T-Flex or FineVision toric implant (about 30/30 and20). So that the groups are comparable, the inclusion and exclusion criteria will be those applicable to a multifocal implant.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
To observe the rotational stability of the implant | 6 Months
  Observation of rotational stability of the implant

SECONDARY OUTCOMES:
Visual Acuity | 6 Months
  To assess the visual acuities with and without correction and the best refraction to assess the benefit of the implants

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Vandekerckhove, MD, Principal Investigator — Vista Alpina Eye Cente, Visp, Switzerland, 3930
Locations (1):
- Vista Alpina Eye Center, Visp, Switzerland